CLINICAL TRIAL: NCT00015860
Title: A Phase I/II Trial of STI-571 and Chemotherapy in Lymphoid Blast Crisis of Chronic Myeloid Leukemia and Philadelphia Chromosome-Positive Acute Lymphoid Leukemia
Brief Title: STI571 Plus Combination Chemotherapy in Treating Patients With Chronic Myelogenous Leukemia or Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068444; UCLA-0011010; UCLA-NCI-4292; NCI-4292
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2003-09

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — Daunorubicin; Imatinib Mesylate; Prednisone; Vincristine

INTERVENTIONS:
Drug: daunorubicin hydrochloride
Drug: imatinib mesylate
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. STI571 may stop the growth of leukemia cells. Combining chemotherapy and STI571 may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy plus STI571 in treating patients who have chronic myelogenous leukemia or acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of daunorubicin when combined with imatinib mesylate, vincristine, and prednisone in patients with lymphoid blastic phase chronic myelogenous leukemia or Philadelphia chromosome-positive acute lymphoblastic leukemia.
* Determine the safety of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the frequency of hematologic and cytogenetic responses in patients treated with this regimen.
* Determine the duration of response of this patient population treated with this regimen.
* Determine the survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of daunorubicin.

Patients who have not previously received imatinib mesylate receive oral imatinib mesylate on days 1-35. Patients who have previously received imatinib mesylate for at least 28 days receive oral imatinib mesylate on days 22-35. All patients receive daunorubicin IV over 2-3 minutes on days 1-3, vincristine IV over 1 minute on days 1, 8, 15, and 22, and oral prednisone on days 1-28. Patients with more than 5% residual blasts in bone marrow on day 28 receive a second course in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of daunorubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the recommended phase II dose.

PROJECTED ACCRUAL: A maximum of 46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Chronic myelogenous leukemia in lymphoid blast crisis
  * Acute lymphoblastic leukemia (ALL) that is in first relapse or failed induction

    * No more than 1 prior course of induction chemotherapy
    * Philadelphia chromosome-positive (Ph+) by cytogenetic analysis OR bcr/abl translocation by fluorescent in situ hybridization
* At least 30% blasts in bone marrow
* Ineligible for or refused allogeneic stem cell transplantation
* Not previously treated with imatinib mesylate OR currently receiving imatinib mesylate with stable disease on 2 bone marrow biopsies at least 2 weeks apart

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin less than 3 times upper limit of normal (ULN)
* ALT and AST less than 3 times ULN

Renal:

* Creatinine less than 2 times ULN

Cardiovascular:

* No New York Heart Association class III or IV cardiac disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 2 weeks after study for female patients and at least 3 months after study for male patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior allogeneic bone marrow or peripheral blood stem cell transplantation
* At least 48 hours since prior interferon alfa

Chemotherapy:

* See Disease Characteristics
* At least 24 hours since prior hydroxyurea
* At least 6 weeks since prior busulfan
* Concurrent hydroxyurea or anagrelide for severe leukocytosis or thrombocytosis allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior therapy for blast crisis except hydroxyurea
* No prior salvage or reinduction therapy for Ph+ ALL
* At least 4 weeks since other prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Paquette, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Oregon Cancer Institute, Portland, Oregon
  - University of Texas - MD Anderson Cancer Center, Houston, Texas